CLINICAL TRIAL: NCT06338774
Title: Targeting Cognitive Control to Improve Physical Activity Adherence in Midlife for Alzheimer's Risk Reduction
Brief Title: Cognitive Control to Boost Physical Activity Adherence
Acronym: BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Northeastern University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michelle W. Voss, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 202310129; R33AG078041 (NIH)
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Physical Inactivity
Keywords: health behavior change; physical activity adherence; exercse
MeSH Terms: conditions — Sedentary Behavior | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Intervention Model Description: Six week parallel group intervention, followed by a 12 week exercise program.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Control: Neutral (CC-N) (Experimental): Game-like cognitive training program that they will run themselves at home up to 5 times per week. A game-like experience begins, where the participant is encouraged to earn points and in-game rewards to advance. In this condition, all the stimuli presented are neutral (not emotionally valenced). After each session, the difficulty of the next session is updated.
  Interventions: Behavioral: Cognitive training; Behavioral: Exercise
- Cognitive Control: Emotionally Valenced (CC-E) (Experimental): Game-like cognitive training program that they will run themselves at home up to 5 times per week. A game-like experience begins, where the participant is encouraged to earn points and in-game rewards to advance. In this condition, all the stimuli presented within the tasks are emotionally valenced.
  Interventions: Behavioral: Cognitive training; Behavioral: Exercise
- Casual Games (Active Comparator): Composed of 6 commercially available computer games. It matches the experimental treatment program in overall program use intensity, time-spent attending, delivered rewards, and overall engagement.
  Interventions: Behavioral: Cognitive training; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Cognitive training — Computerized cognitive training completed on any computer or tablet with internet
Behavioral: Exercise — Aerobic exercise intervention with structured exercise sessions prescribed by a study exercise specialist

SUMMARY:
This trial is designed to develop and test the efficacy of cognitive training strategies to improve self-regulatory capacities for middle-aged adults to adopt and sustain a physically active lifestyle. The main questions it aims to answer are:

* Can cognitive training designed to improve cognitive control improve physical activity adherence?
* What are the psychological, physiological, cognitive, and sociodemographic factors that affect the impact of cognitive control on physical activity adherence?

Participants will

* Complete a 6-week home-based, computerized cognitive training program
* Complete a 6-week home-based, aerobic exercise training program with supervision of a health coach and trainer
* Complete a 6-week home-based, aerobic exercise training program prescribed by a health coach and trainer
* Visit the laboratory before and after cognitive training, and before and after physical training, to complete assessments of cognition and aerobic fitness

DETAILED DESCRIPTION:
Participants will first be screened to ensure eligibility for participating in moderate to vigorous intensity exercise based on health history and approval from their primary physician or equivalent.

Participants will then complete pre-testing and a three-phased intervention. Pre-intervention sessions include study screening, cognitive testing, physical activity assessment, and sub-maximal cardiorespiratory fitness testing.

Participants will then be randomized into one of three cognitive training programs for a 6-week cognitive training intervention. The cognitive training program includes 15 hours of progressive adaptive training. Participants complete 30 min of training 5 days a week to complete a dose of 15 hours of cognitive training. A minimum of 10 hours of completed cognitive training is needed to progress to the exercise training program.

Upon completion of cognitive training, participants will complete testing to assess changes in cognitive function, and then be enrolled in a two-phase exercise intervention. The 12-week exercise program includes a first 6-week introductory and fully supervised training program that builds towards meeting the minimum suggested exercise per week for long-term health benefits (150 minutes/week of moderate intensity exercise). Following the first 6 weeks, participants will be prescribed a maintenance program to be completed fully at home with their heart rate monitor from the study team, and with safety monitoring from our exercise specialist.

After completing the second 6-week exercise intervention, participants will again complete the cognitive and cardiorespiratory fitness testing they did during pre-intervention sessions.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40 and 65 years old
* Full-time working status of an average of 35 hrs./week or more
* Scoring as "Low Active" by the short form of the International Physical Activity Questionnaire (IPAQ)
* Eligible to participate in an aerobic exercise intervention based on the Physical Activity Readiness Questionnaire
* Approval from their Primary Care Physician for approval to participate in the prescribed training program
* Corrected vision of 20/40
* Fluent in English to ensure instructions for cognitive assessments and training are understood clearly

Exclusion Criteria:

* Impairments in hearing inhibiting the ability to discuss study instructions or directions
* Visual impairments that prevent the perception of color, or loss of sight in the visual field
* Qualify as "high risk" for exercise-induced adverse events by American College of Sports Medicine criteria will be excluded, which includes known or symptomatic chronic cardiovascular or metabolic disease
* Not fluent in English
* Inability to comply with experimental instructions or access a tablet or computer to complete computerized training
* Previous diagnosis of a neurological or psychiatric condition, including diagnosis with any of the following: major depression, Attention Deficit Disorder or attention-deficit/hyperactivity disorder (ADHD), schizophrenia or bipolar disorder, multiple sclerosis, epilepsy, meningitis, Parkinson's disease, stroke, Transient Ischemic Attack (TIA), or brain aneurysm surgery.
* Previous diagnosis of a heart condition, cardiovascular disease, or a recent cardiovascular event (such as high blood pressure or cholesterol) that would increase the risk for an adverse event in response to vigorous exercise, Chronic obstructive pulmonary disease (COPD), uncontrolled asthma (this includes anyone who has asthma but is not on medication.
* Previous diagnosis of a chronic condition such as cystic fibrosis, unregulated thyroid disorder (this includes anyone with thyroid disease that is not on medication), untreated diabetes, renal or liver disease, heart murmur, arrhythmia, or irregular heartbeat.
* Previous brain surgery or injury associated with concussion or loss of consciousness that required rehabilitation or caregiver assistance to regain function (i.e., dressing/personal hygiene)
* Previous diagnosis of Alzheimer's or related dementias
* Current or previous cancer treatments within the last 6 months
* Pregnant or trying to get pregnant

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Adherence | 6 weeks
  Proportion of moderate to vigorous physical activity achieved while unsupervised.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Psychological and Brain Sciences Building, Iowa City, Iowa
  - Center for Cognitive and Brain Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol and code for analyses will be shared. We are determining the best outlet for this.